CLINICAL TRIAL: NCT05084820
Title: Effects of Action Observation Treatment on Motor Function in Upper Limb of Patients With Chronic Stroke
Brief Title: Action Observation Treatment on Motor Function in Upper Limb of Patients With Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/20/0213 Hira Rehman
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Stroke
Keywords: stroke; action observation treatment
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: each participant will be requested to draw either number one or two from a box.number one refers to group A and number two refers to group B. Group A patients will receive conventional treatment of 40 minutes in total. group B is experimental group , patients will watch videos of 5 common motor tasks that implicit the usage of items to be used for action observation treatment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Action observation treatment (Experimental): Action observation treatment
  Interventions: Combination Product: Action observation treatment
- conventional treatment (Active Comparator): conventional treatment
  Interventions: Combination Product: conventional treatment

INTERVENTIONS:
Combination Product: Action observation treatment — Participants will watch 5 videos of motor tasks; each video is of 30 sec and watch for 4 times (i.e. for 2 minutes). Then patient will execute the motor act, soon after the observation with an affected limb for 2 minutes, with total rest time of 5 minutes for this treatment. Conventional treatment of muscle stretching, strengthening and ROM exercises will be given for 15 minutes including rest. Total treatment time is 40 minutes.
  Arms: Action observation treatment
Combination Product: conventional treatment — conventional treatment of 40 minutes in total will be performed including Stretching (for 8-10 sec with set of 5 repetitions/ session on each side for 3 minutes total with rest), strengthening (weighted bicep curls, side arm raise and open arm movement exercises with set of 5 repetitions/ session for 9 minutes total with rest), Range of motion exercises active and passive with set of 5 repetitions/ session for 3 minutes total with rest and gripping,reaching, grasping exercises (on each side for total 25 minutes including rest) with assistance of physiotherapist
  Arms: conventional treatment

SUMMARY:
To determine the effects of action observation treatment on motor functions in upper limb of patients with chronic stroke

DETAILED DESCRIPTION:
Stroke is one of the major cause of death in Pakistan and also a prime source of disability in older adults.Mirror neuron system depends on motor regions, and its dominant aspect is that,it is activated for implementation of motor activity and also for its observation. This "dual activation" characteristic of mirror neuron helps in improving the observation and execution of different actions.

aim of this study is to determine the effects of action observation treatment on motor function in upper limb of patients with chronic stroke.

An RCT will be conducted on 14 chronic stroke patients from Omar Hospital and Riphah Rehabilitation Centre Lahore. Patients will be randomly allocated into control group (n=7) and Experimental group (n=7) by lottery method. Control group will be given only conventional treatment that included stretching, strengthening, pinching, gripping, reaching and grasping exercises, while Experimental group received conventional treatment and action observation treatment 3 days/ week for 4 weeks. Treatment outcomes will be assessed on Modified Barthel Index and Fugl-Meyer Assessment for upper extremity (FMA-UE)

ELIGIBILITY:
Inclusion Criteria:

* Chronic Stroke patients (with more than 6 months- 4 years) illness
* Patients that were able to communicate and comprehend oral instructions
* Patients with Mini Mental State Examination (MMSE) score more than 24

Exclusion Criteria:

* Patients having psychiatric histories.
* Visual and hearing impaired patients
* Patients with speech impairment
* Patients with arthritic deformities in upper limb (with or without using assistive device)
* Patients with diagnosed mental illness.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
modified barthal index | 40 minutes
  The Modified Barthel Index score was used for practical evaluation in activities of daily living. The MBI comprises of 10 items, 6 out of 10 items scored from 0-2 points, 2 items scored from 0-3 points and other 2 items scored from 0-3 points, giving a highest total score of 20 points.
Fugl-Meyer Assessment test | 40 minutes
  Fugl-Meyer Assessment test for Upper extermity.to assess level of motor impairment and its recovery after treatment. The FMA-UE comprises of 7 times.

CONTACTS AND LOCATIONS:
Overall Officials: zeest hashmi, MS NMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah international university, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mao H, Li Y, Tang L, Chen Y, Ni J, Liu L, Shan C. Effects of mirror neuron system-based training on rehabilitation of stroke patients. Brain Behav. 2020 Aug;10(8):e01729. doi: 10.1002/brb3.1729. Epub 2020 Jul 1. PMID 32608554
- [Background] Keller J, Stetkarova I, Macri V, Kuhn S, Petioky J, Gualeni S, Simmons capital ES, CyrillicD, Arthanat S, Zilber P. Virtual reality-based treatment for regaining upper extremity function induces cortex grey matter changes in persons with acquired brain injury. J Neuroeng Rehabil. 2020 Sep 12;17(1):127. doi: 10.1186/s12984-020-00754-7. PMID 32919473
- [Background] Keci A, Tani K, Xhema J. Role of Rehabilitation in Neural Plasticity. Open Access Maced J Med Sci. 2019 May 14;7(9):1540-1547. doi: 10.3889/oamjms.2019.295. eCollection 2019 May 15. PMID 31198470
- [Background] Habibi-Koolaee M, Shahmoradi L, Niakan Kalhori SR, Ghannadan H, Younesi E. Prevalence of Stroke Risk Factors and Their Distribution Based on Stroke Subtypes in Gorgan: A Retrospective Hospital-Based Study-2015-2016. Neurol Res Int. 2018 Jul 26;2018:2709654. doi: 10.1155/2018/2709654. eCollection 2018. PMID 30147952